CLINICAL TRIAL: NCT02193893
Title: Safety/Efficacy Study for the Biological Treatment of Amyotrophic Lateral Sclerosis With Autologous Stem/Progenitor Cells
Brief Title: Biological Treatment of Amyotrophic Lateral Sclerosis
Acronym: NeuStem-ALS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Milosz Kawa, Principal Investigator: Boguslaw Machalinski, Professor and Chief, Department of General Pathology, Pomeranian Medical University, Pomeranian Medical University Szczecin, Pomeranian Medical University Szczecin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZPO 02; ZPO 02, ALS-BMSC #01 (Other: Department of General Pathology, PMU in Szczecin)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: cell-based therapy; autologous bone marrow-derived stem/progenitor cells; stem cell infusion, stem cell transplantation; biological therapy with neurotrophic factors; bioactive neurotrophic factors
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem/progenitor cells transplantation. (Active Comparator): Intervention: Biological: Cell-based therapeutics Autologous bone marrow-derived stem/progenitor cells will be transplanted intrathecally (via a standard lumbar puncture) into early vs. progressive ALS subjects.
  Interventions: Other: Biological: Cell-based therapeutics
- Standard treatment of ALS (Sham Comparator): Symptomatic treatment of ALS without biologic cell-based treatment
  Interventions: Other: Symptomatic treatment of ALS

INTERVENTIONS:
Other: Biological: Cell-based therapeutics — Human autologous bone marrow-derived stem/progenitor cell transplantation in ALS patients.
  Arms: Stem/progenitor cells transplantation.
Other: Symptomatic treatment of ALS — Symptomatic neurological treatment of ALS
  Arms: Standard treatment of ALS

SUMMARY:
The purpose of this study is to test the safety and effectiveness of an autologous bone marrow-derived stem/progenitor cells infusion in the subjects with diagnosed amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a universally fatal neurodegenerative condition that causes weakness leading to paralysis and death. Life expectancy is less that 5 years. The cause is generally unknown and there is no effective treatment. Patients with ALS typically exhibit a progressive paralysis due to the continued loss of motoneurons. Intraspinal injections of bone marrow mononuclear cells have been able to ameliorate the course of ALS in murine models. The purpose of this prospective, nonrandomized, open label, pilot study is to conduct the investigation of the safety and efficacy of infusion of autologous bone marrow-isolated stem/progenitor cells with different selected phenotypes into the subjects with diagnosed ALS. Especially, this clinical trial is designated to test the therapeutic (pro-regenerative and neuro-protective) functions of different stem/progenitor cell populations able to secrete bioactive neurotrophic factors. All patients enrolled will have a documented history of ALS disease prior to study enrollment. Patients diagnosed as early stage of ALS with the duration of disease less than 6 months and patients diagnosed with advanced stage of ALS disease with duration of 6-12 months will be recruited and allocated based on their disease severity to two treatment groups: Group I - patients of early ALS disease stage and Group II - patients of advanced ALS disease. Next, autologous bone marrow-isolated stem/progenitor cells administration to the cerebrospinal fluid at the site of the spinal cord will be performed. Finally, treatment safety, adverse events and exploratory parameters, including electromyographic (EMG) studies, forced vital capacity (FVC), functional rating scale (FRS) and maximum voluntary isometric contraction-arm (MVIC-arm) evaluation, to establish ALS progression rate will be recorded throughout the duration of the post-treatment follow up period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of the ALS disease before the cell transplantation (diagnose established following the El Escorial criteria for definite ALS)
* good understanding of the protocol and willingness to consent
* patient is mentally intact and psychologically stable
* signed informed consent

Exclusion Criteria:

Concomitant of other systemic disease or diseases:

* inflammation (high protein or lymphocytosis in the CSF), active infections.
* diabetes,
* cardio-vascular disorders,
* cancer,
* autoimmune diseases
* renal failure,
* impaired hepatic function.
* subject is a respiratory dependent.
* subject unwilling or unable to comply with the requirements of the protocol.
* patient has been treated previously with any cellular therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety of autologous bone marrow stem/progenitor cell infusion in enrolled patients | 1 year
  Confirm the safety of autologous bone marrow stem/progenitor cell infusion in enrolled patients by repeated follow-up over one year with clinical and laboratory evaluations.

SECONDARY OUTCOMES:
Efficacy of autologous bone marrow stem/progenitor cell infusion in enrolled patients. | 1 year
  Confirm the efficacy of autologous bone marrow stem/progenitor cell infusion in enrolled patients by repeated follow-up over one year with clinical and laboratory evaluation tests for neurodegeneration processes analysis and general health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Boguslaw Machalinski, MD, PhD, Study Director — Pomeranian Medical University Szczecin; Przemyslaw Nowacki, MD, PhD, Study Chair — Pomeranian Medical University Szczecin
Locations (1):
- Department of Neurology of Pomeranian Medical University in Szczecin, Szczecin, Poland, Poland

REFERENCES:
- [Derived] Pawlukowska W, Baumert B, Golab-Janowska M, Meller A, Machowska-Sempruch K, Welnicka A, Paczkowska E, Rotter I, Machalinski B, Nowacki P. Comparative assessment and monitoring of deterioration of articulatory organs using subjective and objective tools among patients with amyotrophic lateral sclerosis. BMC Neurol. 2019 Oct 19;19(1):241. doi: 10.1186/s12883-019-1484-2. PMID 31629403